CLINICAL TRIAL: NCT02336243
Title: Docosahexaenoic Acid (DHA) Supplementation During Pregnancy to Prevent Deep Placentation Disorders: A Randomized Clinical Trial and a Study of the Molecular Pathways of Abnormal Placentation Prevention
Brief Title: A Randomized Trial of Docosahexaenoic Acid Supplementation During Pregnancy to Prevent Deep Placentation Disorders
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: University of Chile (Other); Laboratorio Gynopharm - CFR (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 13-217; 1141207 (Other Grant/Funding Number: FONDECYT)
Record Dates: First submitted 2014-10-19; First posted 2015-01-12 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-11

CONDITIONS: Premature Birth; Preeclampsia; Fetal Growth Retardation; Stillbirth
Keywords: docosahexaenoic acid; premature birth; placentation disorders; preeclampsia; fetal growth
MeSH Terms: conditions — Premature Birth; Pre-Eclampsia; Fetal Growth Retardation; Stillbirth | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Docosahexaenoic acid (DHA) (Experimental): Docosahexaenoic acid (DHA) 200 mg capsules, 3 capsules by mouth every day, from early gestation until the end of pregnancy
  Interventions: Dietary Supplement: Docosahexaenoic acid (DHA)
- Placebo (Placebo Comparator): Placebo 200 mg capsules, 3 capsules by mouth every day, from early gestation until the end of pregnancy
  Interventions: Dietary Supplement: Placebo (for Docosahexaenoic acid (DHA))

INTERVENTIONS:
Dietary Supplement: Docosahexaenoic acid (DHA) — Docosahexaenoic acid (DHA), 600 mg per day. Each woman will take three DHA capsules per day (200 mg each), as early in gestation as possible and until the end of pregnancy.
  Arms: Docosahexaenoic acid (DHA)
Dietary Supplement: Placebo (for Docosahexaenoic acid (DHA)) — Each women allocated to the placebo group, will receive three placebo capsules per day. The placebo capsules will have same size, aspect and flavor than the DHA capsules.
  Arms: Placebo

SUMMARY:
This study evaluates the effectiveness of maternal supplementation with Docosahexaenoic acid (DHA) early in pregnancy to reduce the incidence of deep placentation disorders: preterm birth, preterm labor, preterm premature rupture of membranes, preeclampsia and fetal growth restriction. Half of the participants in early pregnancy will receive DHA 600 mg per day, while the other half will receive placebo. Investigators will study also the ability of DHA supplementation, early in pregnancy, to enhance invasion and transformation of spiral arteries by trophoblast, as deep placentation indicators.

DETAILED DESCRIPTION:
Introduction: uteroplacental ischemia may cause preterm birth, either due to preterm labor, preterm premature rupture of membranes, or medical indication (in the presence of preeclampsia or fetal growth restriction). Uteroplacental ischemia is the product of defective deep placentation, that is a failure of invasion and transformation of the spiral arteries by the trophoblast. It has been reported that the failure of normal placentation generates a series of clinical abnormalities nowadays called "deep placentation disorders"; they include preeclampsia (PE), fetal growth restriction (FGR), preterm labor (PL), preterm premature rupture of membranes (PPROM), in utero fetal death and placental abruption. Strategies to prevent deep placentation disorders have been just partially effective. Docosahexaenoic acid (DHA) is an essential fatty acid of the family of long chain polyunsaturated fatty acids (LC-PUFAs) or omega-3 fatty acids. Early reports, suggested that a LC-PUFAs rich diet reduces the incidence of deep placentation disorders. Recent randomized controlled trials are inconsistent to show the benefit of DHA supplementation during pregnancy to prevent deep placentation disorders; but most of them showed that DHA supplementation was associated to lower risk of early preterm birth.

Hypothesis: investigators propose that Docosahexaenoic acid (DHA) supplementation, early in pregnancy, reduces the incidence of deep placentation disorders (preterm birth, preterm labor, preterm premature rupture of membranes, preeclampsia and fetal growth restriction), by improving deep placentation physiology: invasion and transformation of spiral arteries by trophoblast.

General Goals: in this proposal investigators aimed to

1. Assess the effectiveness of maternal supplementation with Docosahexaenoic acid (DHA) early in pregnancy to reduce the incidence of deep placentation disorders: preterm birth, preterm labor, preterm premature rupture of membranes, preeclampsia and fetal growth restriction.
2. Study the ability of DHA supplementation, early in pregnancy, to enhance invasion and transformation of spiral arteries by trophoblast, as deep placentation indicators. Methodology: investigators will conduct a randomized, placebo controlled, double blind, clinical trial of maternal supplementation with DHA (Docosahexaenoic acid) to prevent deep placentation disorders. Women will be recruited before 16 weeks of pregnancy from 5 ambulatory centers, 2.400 pregnant women will be assigned to 600 mg DHA per day or placebo. A composite outcome will be the primary outcome of the study. The components of the composite outcome will be: preterm birth < 34+0 weeks gestation; early preeclampsia (<34+0 weeks) and severe fetal growth restriction (lower than the 2 percentile and < 34+0 weeks). Each of the outcomes of the composite outcome and other clinically relevant maternal and fetal outcomes will be evaluated as the secondary outcomes of the study. Clinical samples will be obtained from pregnant women on both groups, including: plasma, trophoblast, placental bed and myometrium, to study changes of deep placentation or defective placentation markers. Trophoblast cell lines will be used to study the effect of DHA on trophoblast function in vitro.

Expected outcome: In the randomized clinical trial, a 50% reduction in the incidence of the composite outcome in the DHA group (4% placebo vs. 2% DHA) is expected. Investigators expect to decrease defective deep placentation (placental bed biopsies) and defective placentation markers in DHA supplemented women. Investigators expect also to demonstrate that DHA enhances trophoblast migration and invasion in vitro and decreases production of inflammatory cytokines and anti-vasculogenic mediators.

Relevance: if the findings are positive, DHA supplementation, early in pregnancy, will become a safe and effective strategy for primary prevention of highly relevant pregnancy diseases, such as preterm birth, preeclampsia and fetal growth restriction.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years old or older at time of consent
* Capability of the subject to comprehend and comply with study requirements
* Live embryo or fetus (documented with positive fetal heart rate prior randomisation)
* Gestational age before 16+0 weeks of pregnancy
* Planning to deliver at Hospital Dr. Sótero del Río, Hospital Padre Hurtado, or Hospital Clínico Universidad Católica de Chile.

Exclusion Criteria:

* Preexisting diabetes mellitus.
* Uterine anatomic malformation (bicornuate, septate uterus).
* Already taking a prenatal supplement with DHA.
* Bleeding disorder in which DHA was contraindicated.
* Anticoagulant therapy.
* Documented history of drug or alcohol abuse.
* Embryo or Fetus with a known mayor abnormality.
* Unable to give written informed consent.
* In the judgment of the investigator, will be unwilling or unable to comply with study protocol.
* Currently participating in another fatty acid trial

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2400 (Estimated)
Dates: Start 2015-05; Primary Completion 2018-03 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Composite outcome: Preterm birth less than 34+0 gestational weeks or preeclampsia before 34+0 gestational weeks or severe fetal growth restrictions early than 34+0 gestational weeks. | 34 weeks of pregnancy
  * Gestational age (first day of the last menstrual period (LMP) or estimated by ultrasound performed before 12+6 weeks of pregnancy).
  * Severe growth restriction defined as birth weight less than the 2nd percentile of population (according to the current national recommended standard).
  * Preeclampsia defined as blood pressure of 140 mm Hg systolic or higher or 90 mm Hg diastolic or higher that occurs after 20 weeks of pregnancy in a woman with previously normal blood pressure and proteinuria (urinary excretion of 0.3 g protein or higher in a 24-hour urine specimen). Or HELLP syndrome (Haemolysis, Elevated, Liver Enzymes, Low Platelets) or superimposed pre-eclampsia, defined as history of pre-existing hypertension (diagnosed pre-pregnancy or before 20+0 weeks' gestation) with new proteinuria. Or Eclampsia, defined as seizures that cannot be attributable to other causes, in a woman with preeclampsia.

SECONDARY OUTCOMES:
Stillbirth | During pregnancy
  Defined as death of the fetus of at least 500 grams birth weight or, if birth weight is unavailable, a gestational age of at least 20+0 weeks of gestation.
Intrauterine growth restriction | At delivery
  Birth weight less than the 10th percentile of the population standard for the gestational age.
Severe intrauterine growth restriction | At birth
  birth weight less than the 2nd percentile of population (according to the current national recommended standard).
Preterm birth | At birth
  Birth < week 37th, < week 32th, < week 28th
Perinatal death | From the 20th gestational week to the 28th day of life
  number of deaths (fetal deaths and neonatal deaths) of babies ≥500 grams, if birth weight is unavailable, a gestational age ≥20+0 weeks, up to 28 completed days after birth.
Neonatal | From birth to the 28th day of life
  Death of a baby that occurred during the first 28 days of life
Respiratory Distress Syndrome (RDS) | Until the 28th day of life
  Defined as requiring assisted ventilation via endotracheal tube or CPAP (Continuous positive airway pressure) or supplemental oxygen greater or equal to 40% all within the first 24 hours of life and for a duration of greater than or equal to 24 hours, and either an x-ray compatible with RDS or surfactant given between the first 2 and 24 hours of life.
Bronchopulmonary Dysplasia (BPD) | Until the 28th day of life
  Defined as requiring oxygen supplementation at 28 days postnatal age
Intraventricular Hemorrhage (IVH) | Until the 28th day of life
  Diagnosed by imaging, categorized by:
  * Grade 1: blood in germinal matrix
  * Grade 2: blood in germinal matrix and extending into ventricles
  * Grade 3: ventricular enlargement
  * Grade 4: intraparenchymal lesion
Proven Early onset Sepsis | Within the first 48 hours of life
  Within first 48hr of life, confirmed by positive blood or cerebrospinal fluid cultures
Necrotizing Enterocolitis | Until the 28th day of life
  Defined as Bell's stage II (definite case of necrotizing enterocolitis) or greater, or perforation of intestine identified by surgery, or at autopsy. (Neu J. Necrotizing enterocolitis: the search for a unifying pathogenic theory leading to prevention. Pediatr Clin North Am 1996; 43(2): 409-32.)
Low birth weight | At birth
  Number of Infants with a birth weight < 1500 grams, number of Infants with a birth weight < 2500 grams
Admitted to Neonatal Intensive Care Unit (NICU) | Until the 28th day of life
Birth biometry | At birth
  Measurement of ponderal index (birth weight/height^3×100), head circumference (cm), Birth weight (grams).
Cesarean section | At delivery
  Number of deliveries by cesarean section
Preeclampsia | From pregnancy to discharge after delivery
  Defined as blood pressure of 140 mm Hg systolic or higher or 90 mm Hg diastolic or higher that occurs after 20 weeks of pregnancy in a woman with previously normal blood pressure and proteinuria, defined as urinary excretion of 0.3 g protein or higher in a 24-hour urine specimen. Or HELLP (Haemolysis, Elevated, Liver Enzymes, Low Platelets) syndrome Or Superimposed pre-eclampsia, defined as history of pre-existing hypertension (diagnosed pre- pregnancy or before 20+0 weeks' gestation) with new proteinuria. Or Eclampsia, defined as seizures that cannot be attributable to other causes, in a woman with preeclampsia.
Gestational Diabetes (GDM) | During pregnancy
  Screening during pregnancy
Premature rupture of membranes | During pregnancy
  Rupture of the amniotic sac before the onset of labor
Maternal Venous Thrombosis | During pregnancy
  Venous Thrombosis confirmed by imaging during pregnancy
Bleeding during pregnancy | During pregnancy
  Genital bleeding diagnosed during pregnancy
Placental Abruptio | During pregnancy
  Prematurely detachment of a normal positioned placenta for the wall of uterus
Postpartum bleeding | Postpartum period
  Estimated bleeding more than 500 ml after vaginal birth or 1000 ml after cesarean section
Postpartum depression | At the 6th postpartum week
  Postpartum Depression defined by the Edinburgh Postnatal Depression Scale (EPDS)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Carvajal, PhD, Principal Investigator — Pontificia Universidad Catolica de Chile; Claudio Vera, MSc, Study Director — Pontificia Universidad Catolica de Chile; Paulina Rojas, MD, Study Director — Pontificia Universidad Catolica de Chile; Paola Casanello, PhD, Study Director — Pontificia Universidad Catolica de Chile; Mauro Parra, MD, Study Director — University of Chile; Christian Figueroa, MD, Study Director — Pontificia Universidad Catolica de Chile; Sergio González, MD, Study Director — Pontificia Universidad Catolica de Chile
Locations (5):
- Chile (5):
  - Centro de Salud Familiar ANCORA Juan Pablo II, Santiago
  - Centro de Salud Familiar ANCORA Madre Teresa de Calcuta, Santiago
  - Centro de Salud Familiar ANCORA San Alberto Hurtado, Santiago
  - Centro Medico Lira 85, Santiago
  - Centro Medico San Joaquin, Santiago